CLINICAL TRIAL: NCT06209996
Title: Lose Little, Live Longer: A Randomised Controlled Feasibility Trial on a Diet-plus-exercise Weight Management Intervention for Overweight Chinese Cancer Survivors
Brief Title: A Weight Management Intervention for Overweight Chinese Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW23-563
Record Dates: First submitted 2023-12-12; First posted 2024-01-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Weight Loss; Overweight and Obesity
MeSH Terms: conditions — Neoplasms; Weight Loss; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This is a 3-arm feasibility trial study with one intervention group, one active control group and one waitlist control group. Computer-generated block randomization sequences will be generated by a statistician who is blinded to the identity of participants prior to the start of the trial. A block randomisation structure with randomly permuted block sizes of 3 and 6 will be used to reduce selection bias and ensure close balance of the numbers in each arm. The serially labelled opaque sealed envelope method will be used for randomisation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, care provider, and outcomes assessor are masked in terms of not knowing to which condition the participants will be randomized until after the completion of the baseline assessment. The outcomes assessor will break the envelope for the next eligible participant indicating if that participant is to be allocated to intervention or active control or waitlist arms.
  The participants are masked in terms of not knowing that the intervention are hypothesized to yield larger effects than the others (i.e. controls).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L4 weight management intervention (Experimental): A weight management intervention, namely Lose Little, Live Longer (L4), is recently developed to assist overweight cancer survivors in weight loss through lifestyle modification including improved dietary quality and enhanced physical activity levels. Its underlying theoretical framework is principally derived from Social Cognitive Theory (SCT), which have been widely used in health behavioural change interventions.
  Interventions: Behavioral: L4 weight management intervention
- Active control (Active Comparator): A video-based intervention is selected as a low-touch alternative with expected benefits beyond a no treatment control. Participants allocated to the active control arm will receive five educational videos designed to promote a balanced diet and reinforce regular physical activity, weekly through instant messaging.
  Interventions: Behavioral: Active control
- Waitlist (No Intervention): Participants allocated to the waitlist control arm will receive a set of pamphlets with generic, knowledge-based dietary and physical activity information. All pamphlets are developed based on the self-management framework. Participants in this arm will be arranged to attend to the L4 intervention upon completion of the study.

INTERVENTIONS:
Behavioral: L4 weight management intervention — he key goals of the intervention are to: (i) teach knowledge of weight loss benefits and health risks of obesity, (ii) offer skill-based dietary and physical activity advice, (iii) develop an achievable weight loss goal and plan, (iv) enhance weight management self-efficacy, (v) provide access to exercise equipment and resources, and (vi) teach strategies for managing cravings. The L4 intervention is a therapist- delivered intervention involving a registered dietitian and a cancer exercise specialist. Participants allocated to the intervention arm will be provided with a schedule to attend the L4 intervention within four weeks post-baseline via phone. They will receive five intervention sessions (120 min each) on a weekly basis, and will be given home-based practices and reading to practice the skills learnt in each session. The intervention sessions will be delivered in a group format with a maximum of 5 individuals per group, which is likely to enhance accountability.
  Arms: L4 weight management intervention
Behavioral: Active control — A video-based intervention is selected as a low-touch alternative with expected benefits beyond a no treatment control. Participants allocated to the active control arm will receive five educational videos designed to promote a balanced diet and reinforce regular physical activity, weekly through instant messaging, and be encouraged to follow the advice covered in the videos. The materials will be developed based on the existing dietary and physical activity guidelines for cancer survivors. Participants in this arm will be arranged to attend to the L4 intervention upon completion of the study.
  Arms: Active control

SUMMARY:
This study aims to conduct a feasibility trial to examine the feasibility and acceptability of conducting a randomized controlled trial that evaluates the effect of the weight management intervention on anthropometric measures (body weight and BMI), dietary quality, physical activity levels, physical and psychosocial functioning, self- efficacy for weight loss and quality of life.

DETAILED DESCRIPTION:
The primary aim of the proposed study is to assess the feasibility and acceptability of conducting a randomized controlled trial (RCT) that evaluates an adaptive weight management intervention, tailored to Chinese cancer survivors with overweight/obesity after the completion of cancer survivorship care, to improve anthropometric measures (body weight and BMI), dietary quality, physical activity levels, physical and psychosocial functioning, self-efficacy for weight loss and quality of life. According to the Consolidation Standards of Reporting Trials (CONSORT) guidelines for reporting feasibility trials, hypothesis setting for a feasibility trial is not recommended, given that pilot trials are often underpowered to detect difference which instead should be the aim of the main trial.

ELIGIBILITY:
Inclusion Criteria:

* Chinese cancer survivors attending the one-off face-to-face survivorship care clinic
* who are Cantonese- or Mandarin- speaking
* aged 18 or above
* diagnosed with early-stage disease (stage 0-II)
* have completed primary and adjuvant treatments such as chemotherapy and radiotherapy
* and with a BMI ≥ 23 kg/m2, as indicative as overweight or obesity using Asia-Pacific BMI cutoffs at 3-months reassessment

Exclusion Criteria:

* Non-Chinese survivors with advanced or metastatic disease
* who have communication difficulties, mobility impairment or cognitive disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of subject recruitment | baseline
  number of participants consent and being randomized/number of eligible patients x 100
Rate of subject retention | baseline, 3-months and 6- months post-intervention
  number of participants who complete follow-up assessments at 3 and 6 months post-baseline/number of participants enrolled x 100
Adherence rate to intervention | immediate post-intervention
  number of participants who complete the intervention/number of being allocated to attend the intervention x 100
Rate of missing data | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  number of participants with completed datasets for outcome measures/number of participant enrolled x 100
Change of weight | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  Weight will be assessed in light clothing and without shoes using a high-quality segmental body composition monitor (Tanita InnerScan BC545N). To minimise measurement error, weight will be measured twice with accepted values within 0.1kg. If either measure falls outside the accepted range, a third measure will be taken. The average of the two acceptable measures will be used in the analysis.
Change of BMI | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  BMI will be assessed in light clothing and without shoes using a high-quality segmental body composition monitor (Tanita InnerScan BC545N). For the calculation of BMI (kg/m2), height will be measured to 0.01cm using a portable calibrated stadiometer (SECA Stadiometer). To minimise measurement error, weight and height will be measured twice with accepted values within 0.1kg and 0.3cm, respectively. If either measure falls outside the accepted range, a third measure will be taken. The average of the two acceptable measures will be used in the analysis.
change of Self efficacy | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  Self-efficacy for weight loss will be assessed using the 11-item Physical Activity and Nutrition Self-Efficacy (PANSE) scale. Each item is rated on a 9-point Likert scale ranging from 1 "not at all confident" to 9 "highly confident". Total score range is 11 to 99, with higher scores indicative as greater perceived self-efficacy for weight loss. The PANSE has demonstrated strong internal consistency (Cronbach α = .89), convergent validity, and test-retest reliability.(18)

SECONDARY OUTCOMES:
Change of dietary assessment | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  Dietary quality will be assessed with a three-day dietary record. Participants will be instructed to record their diet for three consecutive days including two weekdays and one weekend day, and not to alter their diet deliberately. All dietary records will be coded for the following food groups: (1) total grains, (2) refined grains, (3) whole grains, (4) fruits, (5) vegetables, (6) pork, (7) beef and other red meats, and (8) processed meats.
change of skin carotenoid status | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  Skin carotenoid status, a biomarker of fruit and vegetable intake, will be measured by the Veggie Meter. The Veggie Meter is a non-invasive tool that utilizes the optical method of reflective spectroscopy upon pressure of the fingertip on the lens to measure skin carotenoid status. Three consecutive measurements will be taken per participant without removing the finger from the lens, and the average of the three ranging from 0-800 will be used with higher scores indicating higher fruit and vegetable intake.
Change of physical activity level | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  Physical activity level will be assessed using the Global Physical Activity Questionnaire (GPAQ) developed by World Health Organization. The GPAQ measures how many days per week (0-7 days) and how many times in minutes per day (0-1440 minutes) spent doing different types of physical activity.
change of health-related quality of life | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  The generic EuroQol 5 Dimension 5 Level (EQ-5D-5L) questionnaire evaluates five dimensions including mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each dimension is rated on a 5-level scale (1 = no problem; 2 = slight problem; 3 = moderate problem; 4 = severe problem; 5 = extreme problem).
change of Cancer-specific quality of life | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  Cancer-specific quality of life will be assessed using the standard Chinese version of the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ-C30), which measures five function domains (physical, role, emotional, cognitive and social), three symptom scales (fatigue, pain, and nausea/vomiting), a global health QoL subscale, five single symptoms items (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and financial difficulties, using a 4-point Likert scale ranging from 0 "Not at all" to 3 "Very much"
change of physical and psychological symptom distress | baseline, immediate post-intervention, 3-months and 6- months post-intervention
  Physical and psychological symptom distress will be measured using the 10-item Edmonton Symptom Checklist (ESAS).The ESAS comprises 10 symptoms commonly observed in cancer patients (including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath, and sleep difficulty) that assess three components: physical, emotional and total symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Ng, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- The University of Hong Kong Jockey Club Institute of Cancer Care, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.